CLINICAL TRIAL: NCT06085183
Title: An Open-Label, Randomized, Parallel Group Study to Investigate the Influence of Renal Impairment on the Efficacy and Safety of Two Doses of Bludigo™ When Used as an Aid in the Determination of Ureteral Patency
Brief Title: Indigotindisulfonate Sodium as an Aid in Determination of Ureteral Patency in Patient's With Renal Impairment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prove pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: PVP-22IC05
Record Dates: First submitted 2023-10-06; First posted 2023-10-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ureter Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saline (Placebo Comparator): 48 subjects treated with 5 ml of saline then crossover to treatment arm
  Interventions: Other: Saline Injection 0.9%
- High Dose (Experimental): 24 subjects randomly treated with 5 mL of drug
  Interventions: Other: Saline Injection 0.9%; Drug: Indigotindisulfonate sodium 0.8%
- Low Dose (Experimental): 24 subjects randomly treated with 2.5 mL of drug
  Interventions: Other: Saline Injection 0.9%; Drug: Indigotindisulfonate sodium 0.8%

INTERVENTIONS:
Other: Saline Injection 0.9% — Placebo
Drug: Indigotindisulfonate sodium 0.8% — Experimental contrast dye that is commonly used as a visualization aid in pelvic and abdominal surgeries and for various diagnostic procedures in medical practice.
  Other Names: Bludigo
  Arms: High Dose; Low Dose

SUMMARY:
This is an open label, randomized, multicenter study to evaluate the efficacy and safety of two dose levels (2.5 mL and 5.0 mL) of Indigotindisulfonate Sodium Injection, USP 0.8% when used as an aid in the determination of ureteral patency in patients with different degrees of renal impairment.

DETAILED DESCRIPTION:
An estimated glomerular filtration rate (eGFR) at baseline will be determined using the Modification of Diet in Renal Disease (MDRD) and standardized by using individual's body surface area as described in the FDA's Renal Impairment guidance. Qualified subjects/patients will be stratified into 4 cohorts based on their eGFR at baseline: patients with normal renal function (eGFR ≥ 90 mL/min), patients with mild (eGFR 60-89 mL/min), moderate (eGFR 30-59 mL/min) and severe (eGFR 15-29 mL/min) renal impairment.

Up to ten study centers in the United States will enroll up to approximately 12 subjects per cohort (48 subjects in total) scheduled for a surgical procedure in which the patency of the ureter must be assessed by cystoscopy following the procedure, age 18 to 85 years inclusive covering the full renal function range from normal, mild, moderate, and severe renal impairment. For each subject/patient the study will consist of a screening period (Day -30 to Day -2), a baseline evaluation (Day -1 to Day 1) and a single treatment period (Day 1) with an onsite observation period of 24 hours post-dose. After signing the informed consent, review of inclusion and exclusion criteria will be performed, the collection of concomitant medications, medical history, physical examination, baseline laboratory testing, 12-lead ECG, and vital sign measurements will be completed during the screening visit.

On the day of surgery (Day 1) subjects will be evaluated for eligibility for randomization. Eligible subjects will be stratified by cohort and randomized in a 1:1 ratio to receive a dose of either Bludigo™ high dose (5.0 mL) or Bludigo™ low dose (2.5 mL). All randomized subjects will serve as his/her own control (i.e., intra-patient controlled) for efficacy by receiving a dose of normal saline prior to receiving the randomized Bludigo™ dose. The surgeon will be blinded to the Bludigo™ dose a subject receives. Time of injection of saline and Bludigo™ will be captured.

All treated subjects will have a follow-up visit 7 to 30 days (± 2 days) after the procedure. A final telephone follow-up call will occur on Day 30 (± 2 days) in subjects who have the follow-up visit before Day 28.

Safety assessments will include monitoring of AEs during and post the procedure, clinical laboratory tests, 12-Lead ECG, and vital sign measurements.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between ≥ 18 and ≤ 85 years old
* Subjects who signed a written IRB approved, informed consent form
* Subjects scheduled for a surgical procedure in which the patency of the ureter must be assessed by cystoscopy following the procedure.
* An estimated glomerular filtration rate (eGFR) at baseline will be determined using the Modification of Diet in Renal Disease formula (MDRD) and standardized by using individual's body surface area.

Subject's renal function will be defined based on the following criteria:

* Normal subjects: eGFR of ≥90 mL/min
* Mild renal impairment: eGFR 60 to 89 mL/min
* Moderate renal impairment: eGFR 30 to 59 mL/min
* Severe renal impairment: eGFR 15 to 29 mL/min

Subjects with normal renal function that are judged to be in good health based on medical history, physical examination, vital signs, and laboratory safety tests performed at the Screening Visit and/or prior to administration of study drug.

Patients with renal impairment (mild, moderate, or severe) who have a diagnosis of chronic (>6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in renal function) renal insufficiency meeting criteria at the Screening Visit

Exclusion Criteria:

* Subjects with eGFR <15 mL/min or expected need for dialysis in the near future, or having only 1 kidney
* Subjects with known severe hypersensitivity reactions to Bludigo™ or other dyes, including contrast dyes
* Known history of drug or alcohol abuse within 6 months prior to the time of screening visit
* Subjects, as assessed by the Investigator, with conditions/concomitant diseases precluding their safe participation in this study (e.g., major systemic diseases)
* Unable to meet specific protocol requirements (e.g., scheduled visits) or subject is uncooperative or has a condition that could lead to non-compliance with the study procedures
* Subject is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Subjects with life expectancy < 6 months
* Requirement for concomitant treatment that could bias primary evaluation.
* Subjects who are pregnant or breast-feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Paired sample difference (Bludigo - Saline) in urine jet conspicuity score. | 10 to 15 minutes post study drug administration
  Visualization will be measured by a conspicuity scale designed to provide an objective tool applicable to the visualization of the urinary flow from the ureteral orifices when determining ureter patency. The conspicuity of the urine flow from the ureteral orifices is defined using the 5-point conspicuity score as follows:
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
  Paired sample difference (Bludigo™-Saline) in conspicuity score (PSDCS). PSDCS will be calculated for each ureter (left or right) for each subject from each reviewer.
Responders to Bludigo | 10 to 15 minutes post study drug administration
  Visualization will be measured by a conspicuity scale designed to provide an objective tool applicable to the visualization of the urinary flow from the ureteral orifices when determining ureter patency. The conspicuity of the urine flow from the ureteral orifices is defined using the 5-point conspicuity score as follows:
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
  A subject is considered a responder to Bludigo™ if there is >=1 point improvement in the conspicuity score following the Bludigo™- treatment vs the saline treatment and the conspicuity score for the Bludigo™ treatment must be (3, 4, or 5). The responder criteria will be assessed separately for each ureter (left or right) from each reviewer.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events. | 30 days post study drug administration
  Percentage of patients in each treatment group who experience an adverse event post treatment
Changes in clinical safety laboratory values | 30 days post study drug administration
  Proportion of subjects with clinically important changes in clinical safety laboratory tests after treatment
Changes in vital signs post treatment | 30 days post study drug administration
  Proportion of subjects with clinically important changes in vital signs after treatment
Changes in ECG post treatment | 30 days post study drug administration
  Proportion of subjects with clinically important changes in ECGs after treatment
Changes in blood pressure by dose group and Renal Impairment Cohort | 30 days post study drug administration
  Comparison of post treatment changes in blood pressure by dose group and renal impairment cohort (normal renal function, mild, moderate, and severe impairment)
Changes in heart rate by dose group and Renal Impairment Cohort | 30 days post study drug administration
  Comparison of post treatment changes in heart rate by dose group and renal impairment cohort (normal renal function, mild, moderate, and severe impairment)
Changes in pulse oximetry by dose group and Renal Impairment Cohort | 30 days post study drug administration
  Comparison of post treatment changes in pulse oximetry by dose group and renal impairment cohort (normal renal function, mild, moderate, and severe impairment)
Time to visualization | 10 to 15 minutes post study drug administration
  To describe the time to visualization (TTV) of blue color in the ureteral jets flow following Bludigo™ treatment
Physician Satisfaction | 10 to 15 minutes post study drug administration
  To determine physicians' overall satisfaction with the Bludigo™ treatment by assessing the proportion of surgeons who agree using the 5-point Physician Satisfaction Agreement Scale (PSAS) with the statement:
  "Compared to the saline treatment, my ability to assess ureter patency was improved after the addition of Bludigo™."
  1. = Strongly Agree
  2. = Agree
  3. = Neither Agree nor Disagree
  4. = Disagree
  5. = Strongly Disagree A surgeon's evaluation is considered satisfactory if the rating is either a 1 (strongly agree) or 2 (agree).

OTHER OUTCOMES:
Difference between the Bludigo™ high dose vs Bludigo™ low dose in urine jet conspicuity score | 10 to 15 minutes post study drug administration
  An exploratory comparison will be performed to assess the difference between the Bludigo™ high dose vs Bludigo™ low dose in urine jet conspicuity score.
  The conspicuity of the urine flow from the ureteral orifices is defined using the 5-point conspicuity score as follows:
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
Impact of renal impairment on renal elimination of Bludigo™ | 12 hours post study drug administration
  An exploratory comparison will be performed to assess the impact of renal impairment on renal elimination of Bludigo™.
Urinary excretion of Bludigo in patients with and without renal impairment | 12 hours post study drug administration
  An exploratory assessments of the amount of Bludigo excreted in urine in patients with and without renal impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Boytim, Ph.D., Study Director — Provepharm SAS
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No